CLINICAL TRIAL: NCT02956252
Title: Spinal Versus General Anesthesia for Laparoscopic Cholecystectomy: a Cohort Study With Unselected Consecutive Patients
Brief Title: Spinal Versus General Anesthesia for Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Medical Park Gaziantep Hospital (Other)
Collaborators: Zeugma Saglik Hizmetleri San. Tic. Ltd. Sti. (Industry)
Responsible Party: Principal Investigator, Mehmet Kaplan, Principal Investigator, Medical Park Gaziantep Hospital
Other Study IDs: MK-011-LC
Record Dates: First submitted 2016-10-30; First posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Cholecystitis; Gallbladder Diseases
Keywords: cholecystectomy, laparoscopic; spinal anesthesia; general anesthesia; cholecystectomy
MeSH Terms: conditions — Cholecystitis; Gallbladder Diseases | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Spinal anesthesia group: patients underwent laparoscopic cholecystectomy under spinal anesthesia
  Interventions: Procedure: Spinal anesthesia
- General anesthesia: Patients underwent laparoscopic cholecystectomy under general anesthesia
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Spinal anesthesia — Spinal anesthesia was used in patients who underwent LC
  Groups: Spinal anesthesia group
Procedure: General anesthesia — General anesthesia was used in patients who underwent LC
  Groups: General anesthesia

SUMMARY:
The aim of this study is to compare early postoperative outcomes of unselected consecutive patients underwent laparoscopic cholecystectomy (LC) under spinal versus general anesthesia.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is the gold standard surgical treatment of symptomatic cholecystectomy which traditionally performed under general anesthesia. Laparoscopy has provided many advantages over open surgery for the patients; however, general anesthesia adversely affects patients' early postoperative quality of life (POQoL).

Spinal anesthesia which is a less invasive technique compared to general anesthesia has many advantages regarding the POQoL such as no need to wait for recovery from anesthesia, less nausea and vomiting, less or no pain at the end of surgery, no discomfort associated with intubation, early ambulation, fully awaken and oriented patient in the bed, and less anxious relatives.

LC has been shown to be feasible under spinal anesthesia if performed with proper technique. There are many reports demonstrated the effectiveness and safety of LC under spinal anesthesia in selected patients. However, patients with complicated gallstone disease such as acute, gangrenous or subacute cholecystitis have been considered as unfit cases for LC under spinal anesthesia because of technical difficulties. On the other hand, spinal anesthesia has also been regarded as inappropriate for patients complying with American society for anesthesiology (ASA) III and IV due to the uncontrolled anesthesia risks.

The aim of this study is to compare early postoperative outcomes of unselected consecutive patients underwent LC under spinal versus general anesthesia. If proportion of general anesthesia (PGA) / proportion of spinal anesthesia (PSA) denotes the proportion rate of outcomes in the general anesthesia group (GaG) / spinal anesthesia group (SaG), then two-sided test problem is assessed as follow:

1. Null hypothesis: H0: PGA = PSA. There is no difference between the two anesthesia techniques in terms of primary outcomes.
2. Null hypothesis: H1: PGA ≠ PSA There is a difference between the two anesthesia techniques in terms of primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent laparoscopic cholecystectomy for symptomatic gallstone disease with no restriction for age, gender, ethnicity, disease severity, and ASA grade.

Exclusion Criteria:

* Patients were excluded if they underwent concurrent surgeries, had malignancy suspicion, received or converted to open surgery, and patients who were under spinal anesthesia converted to general anesthesia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between June 2008 and June 2016, all consecutive patients who were admitted or referred to the Medical Park Gaziantep Hospital and underwent LC for symptomatic gallbladder disease were included in the study
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2008-06; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in pain level for the first day | from baseline to postoperative 1, 2, 4 and 6 hours
  Numerical rating scale (NRS) was used
Change in pain level for the first month | From postoperative 1 week to 1 month
  Numerical rating scale was used

SECONDARY OUTCOMES:
Complications | within the postoperative 1 month
  All types of complications were assessed
Mortality | within the postoperative 1 month
  all causes of mortality were recorded
Gastrointestinal quality of life index | change from baseline to postoperative 1 week and 1 month
  A standard form was used under the supervision of experienced independent personal
Patient satisfaction | at postoperative 1 month
  a verbal or visual scale was used

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, M.D., Principal Investigator — Bahcesehir University, BAU

IPD SHARING:
Plan to Share IPD: No